CLINICAL TRIAL: NCT04984707
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study in Healthy Male Subjects With Androgenetic Alopecia to Evaluate the Safety, Tolerability and Pharmacokinetics of KX-826 Following Topical Single Ascending Dose Administration
Brief Title: Safety, Tolerability and Pharmacokinetics of KX826 in Healthy Male Subjects With Androgenetic Alopecia Following Topical Single Ascending Dose Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KX0826-US-1001
Record Dates: First submitted 2021-07-19; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group -KX0826 (Experimental): KX0826 is tropically applied to the scalp of healthy male subjects with Androgenetic Alopecia with a single dose.The applied dosage cohorts are 3mg, 12mg, 48mg and 96mg.
  Interventions: Drug: KX0826
- Control Group- Placebo (Placebo Comparator): Placebo is tropically applied to the scalp of healthy male subjects with Androgenetic Alopecia with a single dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KX0826 — AR antagonist
  Other Names: Pyrilutamide; KX-826
  Arms: Experimental Group -KX0826
Other: Placebo — Placebo of KX-826
  Arms: Control Group- Placebo

SUMMARY:
The study is a Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Dose Escalation Study in Healthy Male Subjects with Androgenetic Alopecia to Evaluate the Safety, Tolerability and Pharmacokinetics of KX-826 Following Topical Single Ascending Dose Administration

DETAILED DESCRIPTION:
A total of 40 subjects will be evaluated with 32 subjects randomized to receive active drug and 8 subjects randomized to receive placebo in a double-blind fashion (ten subjects in each dose cohort with two subjects randomized to placebo for total of four dose cohorts).Subjects were to be assigned to 1 of the 4 dose levels, 3 mg. 12 mg, 48 mg and 96 mg of KX-826 or placebo to match the active product, administered as a topical application.

ELIGIBILITY:
Inclusion Criteria:

1. Are capable of giving informed consent and complying with study procedures;
2. Are males between the ages of 18 and 60 years, inclusive;
3. Have a clinical diagnosis of AGA;
4. Considered healthy by the PI, based on a detailed medical history, full physical examination, clinical laboratory tests, 12-lead ECG and vital signs;
5. Have normal renal and hepatic function as determined by the screening laboratory results;
6. Nonsmoker, defined as not having smoked or used any form of tobacco in more than 6 months before screening;
7. Body mass index (BMI) of 19.0 to 35.0 kg/m2 inclusive and body weight not less than 50 kg;
8. Willing and able to adhere to study restrictions and to be confined at the clinical research center.

Exclusion Criteria:

1. Clinically significant history of gastrointestinal (GI), cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity;
2. Any visible skin disease, damage or condition at the application site which, in the opinion of the investigator, could compromise subject safety and/or interfere with the evaluation of the test site reaction;
3. Subject has any dermatological disorders of the scalp;
4. Subject has a history of hair transplants, hair weaves;
5. Subject has hypersensitivity to previously prescribed minoxidil or finasteride;
6. Known or suspected malignancy;
7. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBs Ag), or hepatitis C (HCV) antibody;
8. A hospital admission or major surgery within 30 days prior to screening;
9. Participation in any other investigational drug trial within 30 days prior to screening;
10. A history of prescription drug abuse, or illicit drug use within 6 months prior to screening;
11. A history of alcohol abuse according to medical history within 6 months prior to screening;
12. A positive screen for alcohol or drugs of abuse;
13. Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products) or acute loss of blood during the 90 days prior to screening;
14. Use of prescription or over the counter (OTC) medications, and herbal (including St John's Wort, herbal teas, garlic extracts) within 14 days prior to dosing (Note: Use of acetaminophen at < 3g/day was permitted until 24 hours prior to dosing);
15. An unwillingness of male participants to use appropriate contraceptive measures if engaging in sexual intercourse with a female partner of childbearing potential. Appropriate measures include use of a condom and spermicide and, for female partners, use of an intrauterine device (IUD), diaphragm with spermicide, oral contraceptives, injectable progesterone, progesterone subdermal implants, or a tubal ligation.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAE) by skin irritation assessments | 3 days
  Skin irritation assessments will be performed during the treatment period. The dermal response score will be based on a visual irritation scale (0-7) that rates the degree of erythema, edema and other signs of cutaneous irritation.
Incidence of treatment-emergent adverse events (TEAE) by vital signs measurements | 3 days
  vital signs (including blood pressure, pulse rate, respiratory rate and oral temperatures)
Incidence of treatment-emergent adverse events (TEAE) by ECG assessment | 3 days
  12-lead ECG
Incidence of treatment-emergent adverse events (TEAE) by clinical lab tests | 3 days
  hematology (hemoglobin, hematocrit, platelet count, RBC count, WBC count, with differential), blood chemistry (BUN, creatinine, total bilirubin, alkaline phosphatase, AST, ALT, GGT, LDH, glucose, albumin, total protein, bicarbonate, phosphate, sodium, potassium, chloride, calcium, total cholesterol, uric acid) and urinalysis (pH, specific gravity, protein, glucose, ketones, bilirubin, blood, nitrites, leukocytes, urobilinogen, microscopic urine analysis on abnormal findings)
Incidence of study drug related TEAEs | 3 days
  incidence of study drug related TEAEs (possibly, probably or definitely)

SECONDARY OUTCOMES:
AUC from time 0 and extrapolated to infinite time, total exposure(AUCinf) | 48 hours
  Pharmacokinetics
AUC from time 0 to the last non-zero concentration(AUClast) | 48 hours
  Pharmacokinetics
Maximum observed concentration (Cmax) | 48 hours
  Pharmacokinetics
Time at which Cmax was first observed(Tmax) | 48 hours
  Pharmacokinetics
half life（T½） | 48 hours
  Pharmacokinetics
Apparent total systemic clearance, calculated as Dose/AUCinf(Cl/F) | 48 hours
  Pharmacokinetics
Apparent volume of distribution(Vd/F) | 48 hours
  Pharmacokinetics
elimination rate constant（Kel） | 48 hours
  Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: David J Wyatt, MD, Principal Investigator — inVentiv Health Clinical Research Services,LLC
Locations (1):
- inVentiv Health Clinical Research Services LLC, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No